CLINICAL TRIAL: NCT04587609
Title: Comparative Effectiveness of Behavioral Interventions, Safety Devices, and Financial Incentives to Reduce Cellphone Use While Driving Among UBI Policy Holders
Brief Title: Reducing Cell Phone Use While Driving Among High Risk UBI Auto Policy Holders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Progressive Auto Insurance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 842968
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Distracted Driving; Driving Impaired
Keywords: financial incentives; gamification; habit formation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control - Standard UBI (No Intervention): Participants will continue to be monitored as a part of their standard UBI and receive educational material about distracted driving in the enrollment period
- Free Phone mount (Other): Participants in this arm will be monitored through standard UBI, receive educational material about distracted driving in the enrollment period, and free phone mounts
  Interventions: Behavioral: Free Phone Mounts
- Commitment + Habit tips (Other): Participants in this arm will receive educational material about distracted driving during the enrollment period, be sent a free phone mount with installation instructions, sign a personalized commitment contract to reduce their phone use, set personal phone use reduction goals, and be sent personalized habit tips framed to help them reduce their handheld phone use while driving;
  Interventions: Behavioral: Free Phone Mounts; Behavioral: Commitment Contract; Behavioral: Personalized Habit Tips
- Habit Formation + Social Gamification (Other): Participants in this arm will will receive all treatments assigned to arm 3, plus social gamification feedback, where each week participants are told if they've reach their weekly handheld phone use while driving reduction goal, and receive or lose points based on whether or not they met their goal. Based on their points participants can either move up or down a level. Each week the participants will also be sent a leader board of their ranking within their group.
  Interventions: Behavioral: Free Phone Mounts; Behavioral: Commitment Contract; Behavioral: Personalized Habit Tips; Behavioral: Social Gamification Feedback
- All + Contest Financial Incentive (Other): Participants in this arm will receive all of the treatments of arm 4 plus be entered into a financial incentive contest where they can either finish in the highest level and split the prize money amongst all participants that reached that level, and the safest driver (driver ranked #1 on the leader board of their group) will receive a small weekly financial prize.
  Interventions: Behavioral: Free Phone Mounts; Behavioral: Commitment Contract; Behavioral: Personalized Habit Tips; Behavioral: Social Gamification Feedback; Behavioral: "Contest" Financial Incentives

INTERVENTIONS:
Behavioral: Free Phone Mounts — Participants will receive free phone mounts
  Arms: All + Contest Financial Incentive; Commitment + Habit tips; Free Phone mount; Habit Formation + Social Gamification
Behavioral: Commitment Contract — Participants will develop and sign a personalized commitment contract where they will create their own weekly goals for phone use reduction, and plan potential future obstacles that may hinder them from reaching their goal and how and plan to overcome that obstacle.
  Arms: All + Contest Financial Incentive; Commitment + Habit tips; Habit Formation + Social Gamification
Behavioral: Personalized Habit Tips — Participants will receive weekly habit formation tips by text message. These messages will be tailored to encourage use of phone mounts, setting up do not disturb while driving, and include their personal obstacles and plans they developed to overcome.
  Arms: All + Contest Financial Incentive; Commitment + Habit tips; Habit Formation + Social Gamification
Behavioral: Social Gamification Feedback — Each week of the intervention period, the participant will be notified whether they met their prior week's goal, stayed about the same, or backslid. Participants will all start with 100 points, and can gain/maintain/lose points each week in the intervention period. Levels are as follows:
  Copper: 0-40 points Bronze: 50-80 points Silver: 90-120 points Gold: 130-160 points Platinum: 170-200 points
  Social competition: participants will be placed in groups of 10 based on similarity of baseline phone use. Weekly leaderboard reports will be sent via email, with SMS reminder. In the leaderboard they'll see themselves as "You".
  Arms: All + Contest Financial Incentive; Habit Formation + Social Gamification
Behavioral: "Contest" Financial Incentives — Participants who finish in the platinum level will receive equal share of a prize, or a small amount will be awarded each week over the course of the intervention period to the weekly "Safest Driver" in each of the social competition cohorts.
  Arms: All + Contest Financial Incentive

SUMMARY:
Insurance User Based Insurance (UBI) users will be invited to participate in a randomized control trial where they will be randomized into 1 of 4 arms: (Arm 1) standard UBI, (Arm 2) Standard UBI + Free phone mounts (Arm 3) Commitment + Habit Tips, (Arm 4) Gamification + Social Competition,(Arm 5) Contest Financial Incentives. Each successive arm will experience all of the elements that the lower-numbered arms will.

DETAILED DESCRIPTION:
Insurance company will invite User Based Insurance app users with more than 2 minutes per hours of handheld phone use in their first month of the insurance program to participate in a study to help them reduce their phone use while driving. Email invitations will include max insurance discount amount for the safest drivers in the customer's demographic group receive for not using their phone while in the User based insurance app. Participants that enroll into the study will be randomized to 1 of 4 arms: (Arm 1) standard UBI where they will continue to be monitored and receive educational material about distracted driving in the enrollment period; (Arm 2) Free phone mounts Arm, this arm will be monitored through standard UBI and receive educational material about distracted driving in the enrollment period, and free phone mounts (Arm 3)+ Commitment + Habit tips, this arm will receive educational material about distracted driving during the enrollment period, be sent a free phone mount with installation instructions, sign a personalized commitment contract to reduce their phone use, set personal phone use reduction goals, and be sent personalized habit tips framed to help them reduce their handheld phone use while driving; (Arm 4) will receive all treatments assigned to arm 2, plus social gamification feedback, where each week participants are told if they've reach their weekly handheld phone use while driving reduction goal, and receive or lose points based on whether or not they met their goal. Based on their points participants can either move up or down a level. Each week the participants will also be sent a leader board of their ranking within their group. (Arm 5) will receive all of the treatments of arm 3 plus be entered into a financial incentive contest where they can either finish in the highest level and split the prize money amongst all participants that reached that level, or the safest driver (driver ranked #1 on the leader board of their group) will receive a small weekly financial prize.

ELIGIBILITY:
Inclusion Criteria:

* Progressive Snapshot Users with policy activated within recruitment period AND reducing in a state which phone use while driving is factored into insurance rating at the time of enrollment
* Has email address

Exclusion Criteria:

* Progressive Snapshot Mobile App not updated to enable push notifications
* Baseline phone use must be greater than or equal to 2 min/hour
* Customer's Snapshot Mobile App does not collect trop data with all sensors active
* Customer in Snapshot program for <30 days or more >70 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1668 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Seconds of active handheld phone use per hour of driving, using smartphone hardware sensors collected via Snapshot telematics app installed on phone | 120 days
  Seconds of active handheld phone use per hour of driving, or percentage of active phone use, including tapping, swiping, and typing. This does not include hands-free phone calls or voice texts. Measurements will be collected using the smartphone's internal hardware, such as an accelerometer gyroscope, and more.

CONTACTS AND LOCATIONS:
Overall Officials: Mucio K Delgado, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayashi Y, Russo CT, Wirth O. Texting while driving as impulsive choice: A behavioral economic analysis. Accid Anal Prev. 2015 Oct;83:182-9. doi: 10.1016/j.aap.2015.07.025. Epub 2015 Aug 13. PMID 26280804
- [Background] Asch DA, Rosin R. Engineering Social Incentives for Health. N Engl J Med. 2016 Dec 29;375(26):2511-3. doi: 10.1056/NEJMp1603978. No abstract available. PMID 28029924
- [Background] Kervick AA, Hogan MJ, O'Hora D, Sarma KM. Testing a structural model of young driver willingness to uptake Smartphone Driver Support Systems. Accid Anal Prev. 2015 Oct;83:171-81. doi: 10.1016/j.aap.2015.07.023. Epub 2015 Aug 13. PMID 26277411
- [Background] Klauer SG, Guo F, Simons-Morton BG, Ouimet MC, Lee SE, Dingus TA. Distracted driving and risk of road crashes among novice and experienced drivers. N Engl J Med. 2014 Jan 2;370(1):54-9. doi: 10.1056/NEJMsa1204142. PMID 24382065
- [Background] Loewenstein G, Asch DA, Volpp KG. Behavioral economics holds potential to deliver better results for patients, insurers, and employers. Health Aff (Millwood). 2013 Jul;32(7):1244-50. doi: 10.1377/hlthaff.2012.1163. PMID 23836740
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920